CLINICAL TRIAL: NCT05713695
Title: Rigorous Evaluation of Strategies to Prevent Overdose Through Linking People With Illicit Substance Use Disorder to Recovery Support Services
Brief Title: Supporting Treatment Access and Recovery Through Linkage and Support
Acronym: STAR-LS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); University of Massachusetts, Lowell (Other); University of Massachusetts, Amherst (Other)
Responsible Party: Principal Investigator, David Smelson, Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000749
Record Dates: First submitted 2023-01-27; First posted 2023-02-06 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Mental Health Disorders; Substance Use Disorders
Keywords: Co-Occurring Disorders; Opioid Overdose; Mental Health Disorders; Substance Use; Medication for Opioid Use Disorder (MOUD); Peer Support; Medication Assisted Treatment (MAT); Healthcare Access; Social Determinants of Health; Coordination of Care; Socioecological Model; Multi-component Interventions; Addiction; Equity
MeSH Terms: conditions — Substance-Related Disorders; Opiate Overdose; Behavior, Addictive

STUDY DESIGN:
Intervention Model Description: MISSION is a time-limited, cross disciplinary, team-based wraparound approach that provides 6 months of psychosocial treatment combined with assertive outreach, empowering clients to access and engage in care and community services to promote recovery. The MISSION treatment curriculum integrates 3 evidence-based practices along with MOUD: 1) Critical Time Intervention (CTI), a time-limited form of assertive community treatment; 2) Dual Recovery Therapy (DRT), which is integrated mental health and substance use group therapy; and 3) Peer Support (PS), offering support for people in recovery by people in recovery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Full MISSION (Experimental): Participants assigned to this condition will receive full MISSION services. MISSION services include 6-months of integrated mental health and substance use treatment and treatment planning with the MISSION Case Manager (13 session curriculum) and Peer Support Specialist (11 session curriculum). Content of these sessions will be directed using the MISSION Treatment Manual and Consumer Workbooks. MISSION teams will also provide linkages and supports to treatment services within the participant's community throughout the duration of the study.
  Interventions: Behavioral: Full MISSION
- Linkage Only Delivered by a Peer Specialist (Active Comparator): Our Linkage only arm delivered by a Peer Specialist will act as the comparison group to the MISSION arm. Participants randomized to the linkage only arm will receive 6-months of linkage care from a Peer Specialist. The Peer Specialist will provide informal treatment planning as well as linkages and support to community services, but will not provide integrated dual disorders treatment, nor will this arm utilize any MISSION materials or offer Peer led groups.
  Interventions: Behavioral: Linkage Only Delivered by a Peer Specialist

INTERVENTIONS:
Behavioral: Full MISSION — MISSION is a time-limited, cross disciplinary, team-based wraparound approach that provides 6 months of psychosocial treatment combined with assertive outreach, empowering clients to access and engage in care and community services to promote recovery. The MISSION treatment curriculum integrates 3 evidence-based practices: 1) Critical Time Intervention (CTI), a time-limited form of assertive community treatment; 2) Dual Recovery Therapy (DRT), which is integrated mental health and substance use group therapy; and 3) Peer Support (PS), offering support for people in recovery by people in recovery.
  Arms: Full MISSION
Behavioral: Linkage Only Delivered by a Peer Specialist — Linkage only is provided via Peer Specialists whom have lived experiences similar to that of our participants. Linkage only includes informal treatment planning and linkages and supports to needed community services.
  Arms: Linkage Only Delivered by a Peer Specialist

SUMMARY:
This 3-year Hybrid Type 1 study will randomize 208 people with co-occurring substance use and mental health disorders (COD) referred from the Worcester Hub. This study seeks to evaluate the effectiveness of MISSION, a multi-component team approach, versus linkage with a Peer Specialist on improving outcomes among individuals with CODs. We expect that individuals receiving MISSION versus linkage only will show greater improvement in treatment engagement, substance use, and mental health outcomes. This study will also concurrently conduct a process evaluation to inform sustainability and future implementation of such interventions.

DETAILED DESCRIPTION:
Addiction is a growing public health problem in the United States (U.S.), with nearly 21 million Americans meeting criteria for substance use disorder (SUD), 1.6 million meeting criteria for opioid use disorder (OUD), and opioid-related overdoses have increased by 50% over the past 5 years. Among people with SUD, 49% have comorbid mental health disorders (COD). Individuals with COD are vulnerable to substance use relapses, mental illness exacerbations, overdoses, homelessness, and criminal justice involvement. However, despite the high rates of morbidity, mortality, and broad social determinant of health needs among people with COD, only 8% of individuals in the U.S. received treatment for both mental illness and SUD. Among those with a COD receiving treatment, 6-month engagement rates are as low as 16% for psychosocial treatments, and 90% of individuals leaving treatment will relapse within 12 weeks. Massachusetts is also hard hit, with a 16% higher SUD prevalence compared to the U.S., and Worcester, the second largest city in Massachusetts, is disproportionately affected by SUD, having one of the highest overdose rates in the state and is ranked 2nd on the Center for Disease Control and Prevention's social vulnerability index. These findings highlight the need to improve treatment access and engagement to support recovery in Worcester, Massachusetts. Both linkage and multicomponent wraparound models have gained popularity as a solution to increase treatment access and engagement. Maintaining Independence and Sobriety through Systems Integration, Outreach and Networking (MISSION) is a hybrid multicomponent linkage and treatment approach, providing assertive outreach linkage support combined with psychosocial treatment, delivered by a cross disciplinary team. MISSION is aligned with the Social Ecological Model (SEM) to address multilevel client needs via 3 evidence-based practices. They include 1) Critical Time Intervention (CTI), a time-limited form of assertive community treatment; 2) Dual Recovery Therapy (DRT), which is integrated group therapy for COD; and 3) Peer Support (PS), offering support for people in recovery by people in recovery. In response to Funding Opportunity Announcement (RFA-CE-22-010), the proposed 3-year Hybrid Type I study, "Supporting Treatment Access and Recovery through Linkage and Support (STAR-LS)," will recruit and randomize 208 patients with COD in Worcester, MA in the Hub, a program run by the Worcester Health and Human Services to one of the following conditions: 1) MISSION; or 2) Peer Support (linkage only). There are three specific aims: Aim 1: To evaluate the effectiveness of MISSION or compared to Peer Support to improve engagement, substance use and mental health symptoms. Aim 2: To examine mechanisms of action of the interventions. Aim 3: To conduct a sequential mixed methods process evaluation to inform sustainability and future implementation. This proposal is aligned with CDC's Strategic Priority Areas and Health People 2030 Core Objectives as it intends to improve behavioral health outcomes strengthen and sustain the recovery ecosystem for people with COD.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 or older;
* Have a COD (1 or more substance use disorders (e.g., alcohol and illicit substances), and a mental health disorder (including depression, anxiety, trauma related disorders, bipolar, and/or schizophrenia);
* Are in the Hub; and
* Are not engaged in other ongoing multi-component treatment for COD with a behavioral health treatment provider or have not seen their provider for at least 3 months.

Exclusion Criteria:

* We will exclude individuals who are acutely psychotic, acutely suicidal with a plan, or homicidal
* Or with concurrent severe alcohol use disorder or high dose benzodiazepine requiring detoxification.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Self-report opioid use and other substance use | Baseline
  Measured by self-report days of use using the Time-line Follow Back (TLFB)
Self-report opioid use and other substance use | 3-months
  Measured by self-report days of use using the Time-line Follow Back (TLFB)
Self-report opioid use and other substance use | 6-months
  Measured by self-report days of use using the Time-line Follow Back (TLFB)
Self-report opioid use and other substance use | 9-months
  Measured by self-report days of use using the Time-line Follow Back (TLFB)
Mental Health Functioning | Baseline
  Measured by self-report mental health symptoms on Behavior and Symptom Identification Scale (BASIS-24)
Mental Health Functioning | 3-months
  Measured by self-report mental health symptoms on Behavior and Symptom Identification Scale (BASIS-24)
Mental Health Functioning | 6-months
  Measured by self-report mental health symptoms on Behavior and Symptom Identification Scale (BASIS-24)
Mental Health Functioning | 9-months
  Measured by self-report mental health symptoms on Behavior and Symptom Identification Scale (BASIS-24)
PTSD Symptoms | Baseline
  Measured by self-report PTSD symptoms on Patient Checklist (PCL-5)
PTSD Symptoms | 3-months
  Measured by self-report PTSD symptoms on Patient Checklist (PCL-5)
PTSD Symptoms | 6-months
  Measured by self-report PTSD symptoms on Patient Checklist (PCL-5)
PTSD Symptoms | 9-months
  Measured by self-report PTSD symptoms on Patient Checklist (PCL-5)
Mental Health Impairment | Baseline
  Measured by self-report on World Health Organization Disability Assessment (WHODAS 2.0)
Mental Health Impairment | 3-months
  Measured by self-report on World Health Organization Disability Assessment (WHODAS 2.0)
Mental Health Impairment | 6-months
  Measured by self-report on World Health Organization Disability Assessment (WHODAS 2.0)
Mental Health Impairment | 9-months
  Measured by self-report on World Health Organization Disability Assessment (WHODAS 2.0)
Psychiatric Severity | Screening
  Measured by Structured Clinical Interview for Diagnostic Statistical Manual (DSM)-5 (SCID-RV)
Psychiatric Severity | Baseline
  Measured by Structured Clinical Interview for Diagnostic Statistical Manual (DSM)-5 (SCID-RV)
Psychiatric Severity | 3-months
  Measured by Structured Clinical Interview for Diagnostic Statistical Manual (DSM)-5 (SCID-RV)
Psychiatric Severity | 6-months
  Measured by Structured Clinical Interview for Diagnostic Statistical Manual (DSM)-5 (SCID-RV)
Psychiatric Severity | 9-months
  Measured by Structured Clinical Interview for Diagnostic Statistical Manual (DSM)-5 (SCID-RV)
Health functioning | Baseline
  Measured by the World Health Organization Quality of Life Scale Brief Version (WHOQOL-BREF)
Health functioning | 3-months
  Measured by the World Health Organization Quality of Life Scale Brief Version (WHOQOL-BREF)
Health functioning | 6-months
  Measured by the World Health Organization Quality of Life Scale Brief Version (WHOQOL-BREF)
Health functioning | 9-months
  Measured by the World Health Organization Quality of Life Scale Brief Version (WHOQOL-BREF)
Therapeutic Alliance Client | Baseline
  Measured by Working Alliance Inventory-C
Therapeutic Alliance Client | 3-months
  Measured by Working Alliance Inventory-C
Therapeutic Alliance Client | 6-months
  Measured by Working Alliance Inventory-C
Therapeutic Alliance Client | 9-months
  Measured by Working Alliance Inventory-C
Therapeutic Alliance Therapist | Baseline
  Measured by Working Alliance Inventory-T
Therapeutic Alliance Therapist | 3-months
  Measured by Working Alliance Inventory-T
Therapeutic Alliance Therapist | 6-months
  Measured by Working Alliance Inventory-T
Therapeutic Alliance Therapist | 9-months
  Measured by Working Alliance Inventory-T
Recovery Capital | Baseline
  Measured by Assessment of Recovery Capital (ARC)
Recovery Capital | 3-months
  Measured by Assessment of Recovery Capital (ARC)
Recovery Capital | 6-months
  Measured by Assessment of Recovery Capital (ARC)
Recovery Capital | 9-months
  Measured by Assessment of Recovery Capital (ARC)
Alcohol or other drug 12-Step Participation | Baseline
  Measured by self-report using the Alcoholics Anonymous Inventory (AAI)
Alcohol or other drug 12-Step Participation | 3-months
  Measured by self-report using the Alcoholics Anonymous Inventory (AAI)
Alcohol or other drug 12-Step Participation | 6-months
  Measured by self-report using the Alcoholics Anonymous Inventory (AAI)
Alcohol or other drug 12-Step Participation | 9-months
  Measured by self-report using the Alcoholics Anonymous Inventory (AAI)
Overdose Risk | Baseline
  Self-report using the Overdose Risk Questionnaire (OdRi)
Overdose Risk | 3-months
  Self-report using the Overdose Risk Questionnaire (OdRi)
Overdose Risk | 6-months
  Self-report using the Overdose Risk Questionnaire (OdRi)
Overdose Risk | 9-months
  Self-report using the Overdose Risk Questionnaire (OdRi)
Number of Outreach and Linkage Sessions | Baseline
  Self-reported using the Psychosocial Treatment & Healthcare Services Tracking Sheet
Number of Outreach and Linkage Sessions | 3-months
  Self-reported using the Psychosocial Treatment & Healthcare Services Tracking Sheet
Number of Outreach and Linkage Sessions | 6-months
  Self-reported using the Psychosocial Treatment & Healthcare Services Tracking Sheet
Number of Outreach and Linkage Sessions | 9-months
  Self-reported using the Psychosocial Treatment & Healthcare Services Tracking Sheet
Baseline Demographics | Baseline
  Self-reported using the Addiction Severity Index (ASI)
Suicide Severity | Screening
  Self-report using the Columbia-Suicide Severity Rating Scale (C-SSRS)
Community Health & Social Needs | Baseline
  Self-report using the Accountable Health Communities & Health-Related Social Needs
Fidelity to Intervention | Weekly
  Measured via clinical staff submitting weekly treatment fidelity logs
Acceptability & Appropriateness | 6-months
  Using the The Acceptability of Intervention Measure (AIM) and Intervention Appropriateness Measure (IAM)
Feasibility of Intervention | 6-months
  Using the Feasibility of Intervention Measure (FIM)
Satisfaction with Care | 6-months
  Self-report using the Treatment Satisfaction Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: David Smelson, PsyD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Consistent with Health and Human Services/Center for Disease Control and Prevention (CDC) policy, research resources and data will be made readily available for research purposes to qualified individuals within the scientific community after publication of any scholarly work. Scholarly publications will also be immediately available to the public on PubMed Central. Additionally, raw and analyzed de-identified data used in publications will be responsibly shared through submissions to a CDC-approved data repository. Other methods for data sharing will be via presentations at professional conferences and, as findings permit, disclosure of summary data to professionals and the general public. To the extent feasible and appropriate, we will share pre-publication findings with colleagues who have a demonstrable, legitimate scientific interest that may be addressed by research findings. We expect to further disseminate the study via gray literature and the project website.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: De-identified data will be shared with qualified and approved researchers via an appropriate data repository. Research data will be destroyed 6 years after the end of the Fiscal Year in which the study is completed. The master list of identifiers will be destroyed at the 6-year mark or when all statistical analyses have been completed and scientific papers have been published, whichever comes first.
Access Criteria: We will share findings with colleagues who have a demonstrable, legitimate scientific interest that may be addressed by research findings.